CLINICAL TRIAL: NCT00107120
Title: A Double-blind Flexible Dose Study of Escitalopram in Pediatric Patients With Major Depressive Disorder
Brief Title: The Safety and Efficacy of Escitalopram in Pediatric Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCT-MD-32
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2009-11-04 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Adolescents; Escitalopram; Pediatrics
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Escitalopram (Experimental): Escitalopram 10mg once daily for three weeks, 10-20mg once daily for up to the remaining 5 weeks
  Interventions: Drug: Escitalopram
- 2 (Placebo Comparator): Placebo once daily for up to 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10mg per day for three weeks, 10-20mg per day for up to the remaining 5 weeks
  Other Names: Lexapro (TM)
  Arms: Escitalopram
Drug: Placebo — Placebo once daily for up to 8 weeks
  Arms: 2

SUMMARY:
Depression affects approximately 2.5% of children and 8% of adolescents. Escitalopram is the S-enantiomer of citalopram. Both escitalopram and citalopram are selective serotonin reuptake inhibitors (SSRIs) and are used to treat depression in adults. This study is designed to provide a systematic evaluation of the safety and efficacy of escitalopram in the treatment of depressed pediatric patients, 12 to 17 years of age. Patients completing the study will be eligible to enter an open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) diagnostic criteria for Major Depressive Disorder.
* Patient's current depressive episode must be at least 12 weeks in duration
* Patient must have a parent or caregiver who must agree to accompany the patient to all clinic visits.

Exclusion Criteria:

* Patients who currently meet DSM-IV criteria for:

  1. attention deficit-hyperactivity disorder
  2. obsessive-compulsive disorder
  3. posttraumatic stress disorder
  4. bipolar disorder
  5. pervasive developmental disorder
  6. mental retardation
  7. conduct disorder
  8. oppositional defiant disorder
* Patients who are considered a suicide risk (have active suicidal ideation), who have made a suicide attempt, or who have ever been hospitalized because of a suicide attempt.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2005-03; Primary Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ventura, PhD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (28):
- United States (28):
  - University of California at Davis, MIND Institute, Health Services, Sacramento, California
  - UCSD Outpatient Psychiatry Services, San Diego, California
  - PCSD - Feighner Research, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida - Child Study Program, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Kolin Research Group, Winter Park, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Clinco, Terre Haute, Indiana
  - Psychiatric Associates, Overland, Kansas
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Capitol Clinical Research Associates, Rockville, Maryland
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Creighton University Medical School, Department of Psychiatry, Omaha, Nebraska
  - CNS Research Institute, Clementon, New Jersey
  - Pulmonary and Allergy Associates, P. A., Summit, New Jersey
  - North Carolina Neuropsychiatry, PA, Chapel Hill, North Carolina
  - University of Cincinnati College of Medicine, Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Division of Child & Adolescent Psychiatry, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - University of Pennsylvania, Department of Psychiatry, Mood & Anxiety Disorders Section, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Friends Hospital, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Center for Pediatric Psychiatry, Dallas, Texas
  - University of Texas Medical Branch, Department of Psychiatry & Behavioral Sciences, Galveston, Texas
  - Brighton Research Group, LLC, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Result] Emslie GJ, Ventura D, Korotzer A, Tourkodimitris S. Escitalopram in the treatment of adolescent depression: a randomized placebo-controlled multisite trial. J Am Acad Child Adolesc Psychiatry. 2009 Jul;48(7):721-729. doi: 10.1097/CHI.0b013e3181a2b304. PMID 19465881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from April 1, 2005 through March, 2007 at 40 centers in the US.
Pre-assignment Details: 2 week screening with one-week single-blind placebo. Patients meeting selection criteria at baseline were randomized to once daily escitalopram 10-20mg/day or placebo (1:1).
Groups:
- Escitalopram: Once daily oral administration of escitalopram tablets - 1 tablet (10mg) for the first three weeks, then 1 tablet (10mg or 20mg) depending on therapeutic response and tolerability.
- Placebo: Once daily oral administration of placebo tablets
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 155 (Safety Population defined as all patients who took at least one dose of double-blind study drug) | 157 (Safety Population defined as all patients who took at least one dose of double-blind study drug)
Completed | 126 | 133
Not Completed | 29 | 24
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 5 | 5
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Lost to Follow-up | 8 | 6
Not completed — Pregnancy | 0 | 1
Not completed — moving away from site | 1 | 1
Not completed — death of parent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 155 | 157 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 155 | 157 | 312
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.6) | 14.5 (1.5) | 14.6 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 92 | 184
  Male | 63 | 65 | 128
Region of Enrollment [Number; unit: participants]
  United States | 155 | 157 | 312

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Depression Rating Scale - Revised (CDRS-R) Total Score
Description: Change from baseline to week 8 in Children's Depression Rating Scale total score. The scale measures 17 depressive symptoms, of which 3 are rated 1-5 and 14 are rated 1-7 (1 = no symptom difficulties; 5 or 7 = severe clinically significant difficulties) for a total score range of 17-113.
Time Frame: Baseline to end of week 8
Population: Efficacy analyses used Intent-To-Treat Population, which consisted of all patients who received at least 1 dose of double-blind study drug & who had at least 1 post-baseline assessment of the CDRS-R. LOCF technique was used to impute missing data. 1 escitalopram pt. did not have a post-baseline CDRS-R total score.
Measure: Mean (Standard Error); unit: Change in total score at endpoint
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 154 | 157
Change in total score at endpoint | -22.4 (1.1) | -18.4 (1.1)
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; The null hypothesis is that there is no difference in the Change from Baseline to Week 8 in CDRS-R total score between treatment groups. The power calculation was based on the change from baseline to Week 8 in CDRS-R total score (LOCF approach). Assuming an effect size (treatment group difference relative to standard deviation) of 0.325, a sample size of approximately 150 patients per treatment group was used to provide at least 80% power at a significance level of 0.05 using a two-sided test; Test type: Superiority or Other; p = 0.022, ANCOVA — Two-sided at 5% level of significance p < 0.05 considered significant; The model included study center and treatment as factors and baseline core as covariate; Least Square Means Difference = -3.4, 95% CI [-6.2 to -0.5], Standard Error of Mean 1.458 — Differences are Escitalopram-Placebo

2. Secondary Outcome: Clinical Global Impressions - Improvement
Description: Clinical Global Impressions - Improvement score at the end of week 8. The scale rates improvement or worsening of patient mental health relative to baseline on a scale from 1 (very much improved) to 7 (very much worse).
Time Frame: CGI-I score at the end of Week 8
Population: The Intent-To-Treat Population was used. The Last Observation Carried Forward (LOCF) technique was used to impute missing data.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 154 | 157
Score on scale | 2.2 (0.1) | 2.5 (0.1)
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Missing values were imputed using the LOCF approach; Test type: Superiority or Other; p = 0.008, ANCOVA — Two-sided at 5% level of significance; The model included treatment and center as factors and baseline CGI-Severity score as covariate; Least Square Means Difference = -0.344, 95% CI [-0.595 to 0.092], Standard Error of Mean 0.1128 — Differences are Escitalopram-Placebo

3. Other Pre Specified Outcome: Children's Global Assessment Scale
Description: Change from baseline to week 8 in CGAS score which rates the patient's general level of functioning for the past 14 days on a scale of 1 (most impaired) to 100 (healthiest).
Time Frame: At baseline and end of week 8
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Change in score
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 154 | 157
Change in score | 14.7 (1.0) | 12.4 (1.0)
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; ANCOVA on the Change from Baseline to Week 8 in CGAS score. The model included treatment and center as factors and baseline score as covariate. Missing values were imputed using the LOCF approach; Test type: Superiority or Other; p = 0.103, ANCOVA — Two-sided at 5% level of significance; Least Square Means Difference = 2.169, 95% CI [-0.439 to 4.777], Standard Error of Mean 1.324 — Differences are Escitalopram-Placebo

ADVERSE EVENTS:
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 4/155 | 2/157
Other Adverse Events (participants affected / at risk) | 121/155 | 118/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=155) | Placebo (N=157)
Inflicted Injury (General disorders) | 2 | 0
Irritability (Psychiatric disorders) | 1 | 0
Suicidal Tendency (Psychiatric disorders) | 1 | 1
Depression Aggravated (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=155) | Placebo (N=157)
Headache (Nervous system disorders) | 39 | 40
Insomnia (Psychiatric disorders) | 16 | 10
Nausea (Gastrointestinal disorders) | 16 | 13
Abdominal Pain (Gastrointestinal disorders) | 14 | 11
Inflicted Injury (General disorders) | 14 | 21
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 13 | 15
Fatigue (General disorders) | 12 | 13
Influenza-like Symptoms (General disorders) | 11 | 5
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Menstrual Cramps (Reproductive system and breast disorders) | 10 | 14
Vomiting (Gastrointestinal disorders) | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Upper Respiratory Tract Infections (Respiratory, thoracic and mediastinal disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 90 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential info. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in pub. On sponsor's request, PI shall delay submission for any pub while sponsor files patent apps. If trial is multi-center, PI agrees that first publication shall be a multi-center pub.